CLINICAL TRIAL: NCT04222478
Title: Interest of Auriculotherapy in the Treatment of Xerostomia.
Acronym: AURICULOXERO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018_0101
Record Dates: First submitted 2019-12-31; First posted 2020-01-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Xerostomia
Keywords: Auriculotherapy; Xerostomia; ENT cancer
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real Auriculotherapy (Experimental): Patients benefit from 3 sessions of auriculotherapy with semi-permanent needles on the 6 points according to the "protocol of Alimi" at one month intervals.
  Interventions: Other: Specific auriculotherapy
- Sham Auriculotherapy (Sham Comparator): Patients are treated according to the same scheme as the experimental group but with semi-permanent needles positioned on non-specific points.
  Interventions: Other: Non-specific auriculotherapy

INTERVENTIONS:
Other: Specific auriculotherapy — 3 sessions of auriculotherapy with semi-permanent needles on the 6 points according to the "protocol of Alimi" at one month intervals.
  Arms: Real Auriculotherapy
Other: Non-specific auriculotherapy — 3 sessions of auriculotherapy with semi-permanent needles on non-specific points.
  Arms: Sham Auriculotherapy

SUMMARY:
The aim of the study is to show that auriculotherapy is effective in the treatment of xerostomia

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old;
* Complain about xerostomia after cervical irradiation in the context of ENT cancer;
* End of radiotherapy> 3 months
* Covered by a national healthcare insurance
* Consent form signed.

Non inclusion Criteria:

* Pregnant or breastfeeding women;
* Local counterindication to auriculotherapy;
* With anticoagulant treatment;
* History or existing of hemophilia;
* Valvular prosthesis;
* Ear's pavilion infection;
* Treatment by auriculotherapy or acupuncture in this indication in the previous 12 months;
* Having started in the 48 hours preceding the first auriculotherapy session, any new management of xerostomia and likely to interfere with the study (specific medication and/or complementary therapeutic management);
* Difficulty to comply with the treatment, questionnaires or study protocol;
* Being deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improvement of salivation after 3 month of treatment (Real Auriculotherapy group compared to Sham Auriculotherapy group) | 3 months
  Show that auriculotherapy (treatment of specific points) is effective in the treatment of xerostomia compared to a "sham" treatment (treatment of non-specific points).
  The relative variation of salivary secretion "after treatment" compared to "before treatment" will be judged on the weight of 3 compresses left 5 minutes in the mouth: 2 in front of the openings of Sténon's canal and 1 on the buccal floor (orifice of Wharton's canal).
  Salivary secretion is measured by the weight in grams of the compresses left in the mouth.
  This measurement is performed at inclusion and after 3 months of treatment. The measurement is made with a jeweler-type precision balance.

SECONDARY OUTCOMES:
Assess the effect of auriculotherapy on the subjective improvement of salivation | 3 months
  Specific xerostomia questionnaire at inclusion and 3 months post-treatment (11 questions with 5 response levels (1 = never / 2 = very rarely / 3 = occasionally / 4 = quite often / 5 = very often) to evaluate Xerostomia symptoms).
Assess the effect of auriculotherapy on the subjective improvement of clinical status | 3 months
  Global Patient Change Impression (GPCI) questionnaire at 3 months post-inclusion. This questionnaire evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status.
Assess the effect of auriculotherapy on the dysgeusia, dysphagia, pain or burning sensations | 3 months
  Simple numerical scales from 0 (best score) to 10 (worst score) at inclusion and at 3 months post-treatment.
Assess the effect of auriculotherapy on anxiety and depression | 3 months
  Hospital Anxiety and Depression questionnaire at inclusion and 3 months post-treatment. The HADS consists of 14 items, scored from 0 to 3, with seven questions relating to anxiety and seven questions relating to depression, allowing 2 scores to be obtained. The highest scores indicating more severe symptoms: "normal" cases (0-7 points); doubtful case (8-10 points); certain cases (11-21 points).
Assess the effect of auriculotherapy on quality of life | 3 months
  EuroQoL five Dimension questionnaire at inclusion and 3 months post-treatment. This questionnaire is designed for the patient to judge the impact of his state of health on his quality of life according to 5 dimensions (mobility, personal autonomy, daily activities, pain / discomfort and anxiety / depression). Each item has 3 response levels (1, 2 and 3) and the combination of the five digits will represent the patient's state of health. It is supplemented by a quality of life thermometer graduated from 0 (worst quality of life) to 100 (best quality of life).
Assess the effect of auriculotherapy on the wish to continue treatment | 3 months
  Patient's desire to continue treatment (question to patient - yes/no response)

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (4):
- France (4):
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan, Brest, Brittany Region
  - Hôpital Forcilles, Férolles-Attilly
  - GHP Saint Joseph, Paris
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No